CLINICAL TRIAL: NCT04166552
Title: A Phase IIa, Double-Blind, Randomised, Intracohort Placebo-Controlled, Multicentre Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of EHP-101 in Patients With Diffuse Cutaneous Systemic Sclerosis
Brief Title: Evaluation of Safety, Tolerability and Preliminary Efficacy of EHP-101 in Diffuse Cutaneous Systemic Sclerosis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor ceasing all operations due to company's shut down
Sponsor: Emerald Health Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EHP-101-SS01
Record Dates: First submitted 2019-11-06; First posted 2019-11-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-09

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Scleroderma; Systemic sclerosis; EHP-101 Oral Solution; dcSSc; diffuse; pathological processes; connective tissue disease; skin disease
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Pathologic Processes; Connective Tissue Diseases; Skin Diseases

STUDY DESIGN:
Intervention Model Description: This is a dose escalation double-blind intracohort trial starting with Cohorts 1 and 2 commencing in parallel and then Cohorts 3 and 4 commencing in parallel
Who Masked: Participant, Investigator
Masking Description: Double (intracohort)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- EHP-101 low dose once a day (Experimental)
  Interventions: Drug: Patients will be randomized to receive EHP-101 or Placebo
- EHP-101 low dose twice a day (Experimental)
  Interventions: Drug: Patients will be randomized to receive EHP-101 or Placebo
- EHP-101 high dose once a day (Experimental)
  Interventions: Drug: Patients will be randomized to receive EHP-101 or Placebo
- EHP-101 high dose twice a day (Experimental)
  Interventions: Drug: Patients will be randomized to receive EHP-101 or Placebo

INTERVENTIONS:
Drug: Patients will be randomized to receive EHP-101 or Placebo — EHP-101 or placebo will be taken once a day
  Arms: EHP-101 high dose once a day; EHP-101 low dose once a day
Drug: Patients will be randomized to receive EHP-101 or Placebo — EHP-101 or placebo will be taken twice a day
  Arms: EHP-101 high dose twice a day; EHP-101 low dose twice a day

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of EHP-101 in adult subjects with diffuse cutaneous Systemic Sclerosis (dcSSc).

DETAILED DESCRIPTION:
An interventional, double-blind, randomized, intracohort placebo-controlled design will be used to test safety, tolerability, pharmacokinetics, and preliminary efficacy of EHP-101 in 36 patients ≥ 18 and ≤ 74 years of age with documented dcSSc. There is a screening period of 28 days, 84 days treatment period, and 28 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients male and female ≥18 years and ≤74 years at the time of consent;
* American College of Rheumatology/ European League Against Rheumatism 2013 Criteria for SSc; dcSSc (skin thickening on upper arms, upper legs, or trunk);
* Documented SSc for up to 6 years from the first non-Raynaud's phenomenon with a total mRSS of ≥15;
* No new or increased doses of immunosuppressants medications within 3 months prior to Screening;
* Effective method of contraception for participants and their partners.

Exclusion Criteria:

* Severe or unstable Systemic Sclerosis (SSc) or SSc with end-stage organ failure;
* Patient with FVC <60%;
* History of clinically significant medical condition or concurrent medical therapies that would exclude the patient, preclude participation in the clinical trial, influence response to study product, or interfere with study assessments;
* History of gastrointestinal dysmotility requiring total parenteral nutrition or hospitalization within 6 months before Visit 1;
* Any one of the following values for laboratory tests at screening:

  * Haemoglobin <9 g/dL;
  * Neutrophils <1.0 x 10^9/L;
  * Platelets <75 x 10^9/L;
  * Estimated creatinine clearance <50 mL/min according to the Cockcroft-Gault equation;
  * Serum transaminases >2.0 x upper normal limit;
  * Total bilirubin ≥1.5 x upper limit of normal.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events | Day 113
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments.

SECONDARY OUTCOMES:
Treatment effect of EHP-101 compared to placebo as measured by the American College of Rheumatology composite response index in diffuse cutaneous Systemic Sclerosis | Day 85 and Day 113
  The ACR CRISS exponential algorithm determines the predicted probability of improvement from baseline, incorporating change in modified Rodnan Skin Score (mRSS), Forced Vital Capacity (FVC) % predicted, physician and patient global assessments, and Scleroderma Health Assessment Questionnaire Disability Index (S-HAQ-DI). The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). Subjects are not considered improved (ACR CRISS score = 0) if they develop new: 1) renal crisis; 2) decline in FVC% predicted by 15% (relative) from baseline and confirmed after 1 month; or 3) left ventricular failure (systolic ejection fraction < 45%); or 4) new pulmonary artery hypertension on right heart catheterization requiring treatment.
Treatment effect of EHP-101 compared to placebo in modified Rodnan Skin Score | Day 85 and Day 113
  The mRSS consists of an evaluation of patient's skin thickness rated by clinical palpation using a 0-3 scale (0 = normal skin; 1 = mild thickness; 2 = moderate thickness; 3 = severe thickness with inability to pinch the skin into a fold for each of 17 surface anatomic areas of the body: face, anterior chest, abdomen, and, with right and left sides of the body separately evaluated, the fingers, forearms, upper arms, thighs, lower legs, dorsum of hands and feet. Individual values are summed and defined as the total skin score. Total score is 0 to 51.
Treatment effect of EHP-101 compared to placebo in forced vital capacity percent predicted | Day 85 and Day 113
  Forced vital capacity (FVC) is a standard pulmonary function test used to quantify respiratory muscle weakness . FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%
Treatment effect of EHP-101 compared to placebo in physician global assessment score | Day 85 and Day 113
  The Physician Global Assessment of disease activity will be performed using a segmented numerical version of the visual analogue scale in which the physician selects a whole number (0-10 integers) that best reflects the overall disease activity. The numerical rating score is anchored by 2 verbal descriptors, one of "no disease activity" (score of 0) and one of "worse imaginable disease activity" (score of 10), with numbers 1-9 spaced equidistance in between. The physician will select an integer to describe disease activity. The recall period is one week.
Treatment effect of EHP-101 compared to placebo in patient global assessments score | Day 85 and Day 113
  The Patient Global Assessment will be performed with a segmented numerical version of the visual analogue scale in which the subject selects a whole number (0-10 integers) that best reflects the overall disease activity. The numerical rating score is anchored by two verbal descriptors, one of "no disease activity" (score of 0) and one of "worse imaginable disease activity" (score of 10), with numbers 1-9 spaced equidistance in between. The subject will select an integer to describe disease activity. The recall period is one week.
Treatment effect of EHP-101 compared to placebo in Scleroderma Health Assessment Questionnaire - Disability Index | Day 85 and Day 113
  S-HAQ-DI includes 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are two or three questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). The eight scores of the eight sections are summed and divided by 8. If one section is not completed by a subject, the summed score is divided by 7. As such, maximum scores can vary with a min of 0. The result is the DI, the disability index or functional disability index. The recall period is one week.

OTHER OUTCOMES:
Change from baseline of EHP-101 compared to placebo in Patient-Reported Outcomes Measurement Information system-29 Short | Day 85
  (PROMIS)-29 Short measures self-reported physical, mental wellbeing. It consists of 29 questions. The questions are ranked on a 5-point Likert Scale.
Change from baseline of EHP-101 compared to placebo in 5 dimensions Itch Score | Day 85
  5-D Itch Score comprises the following 5 dimensions: degree, duration, direction, disability and distribution. The recall period is two weeks.
Change from baseline of EHP-101 compared to placebo in University of California, Los Angeles Scleroderma Clinical Trial Consortium Gastrointestinal Tract Questionnaire | Day 85
  The UCLA SCTC GIT 2.0 has 7 multi-item scales: Reflux, Distension/Bloating, Diarrhea, Fecal Soilage, Constipation, Emotional Well-being, and Social Functioning and a total GIT score. All scales are scored from 0 [better health-related quality of life (HRQOL)] to 3 (worse HRQOL) except the diarrhea and constipation scales (ranges 0-2 and 0-2.5, respectively). The Total GIT Score, is developed by averaging 6 of 7 scales (excluding constipation). The recall period is one week.
Change from baseline of EHP-101 compared to placebo in Functional Assessment of Chronic Illness Therapy: Fatigue | Day 85
  The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The composite score of all item will be used. The total score ranges from 0 to 52. The recall period is one week.
Change from baseline of EHP-101 compared to placebo in the European Quality of Life 5 Domain Questionnaire | Day 85
  The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Quantitation of drug plasma levels at different timepoints to determine trough | Day 113
  To determine trough level plasma concentrations of drug substance of EHP 101

CONTACTS AND LOCATIONS:
Locations (23):
- United States (13):
  - Arizona Arthritis & Rheumatology Associates, P.C., Phoenix, Arizona
  - Care Access Research - Huntington, Huntington Beach, California
  - Pacific Arthritis Care Center, Los Angeles, California
  - UCLA Division of Rheumatology, Los Angeles, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Yale University, New Haven, Connecticut
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - Life Clinical Trials, Margate, Florida
  - Novel Clinical Research Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - Footscray Hospital, Footscray
  - Griffith University, Gold Coast
  - Fiona Stanley Hospital, Murdoch
  - Westmead Hospital, Sydney
- Wellington Hospital, Wellington, New Zealand
- Puerto Rico (3):
  - Centro Reumatologico, Caguas
  - Mindful Medical Research, San Juan
  - University of Puerto Rico, Medical Sciences Campus, San Juan

IPD SHARING:
Plan to Share IPD: No